CLINICAL TRIAL: NCT02012504
Title: Antidepressant Monotherapy on Depressive and Anxiety Symptom in Chinese Patients Who Meet Comorbidity of Major Depressive Disorder (MDD) and Generalized Anxiety Disorder (GAD)
Brief Title: Antidepressant Monotherapy on Depressive and Anxiety Symptom in Chinese Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2012-127
Record Dates: First submitted 2013-11-15; First posted 2013-12-16 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Adverse Drug Reaction; Anxiety Disorders and Symptoms
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Western medicine: venlafaxine or escitalopram
- Chinese medcine: Shuganjieyu capsule

SUMMARY:
The primary objective is to evaluate the improvement of antidepressant monotherapy on depressive and anxiety symptom in Chinese patients who meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for the comorbidity of major depressive disorder (MDD) and generalized anxiety disorder (GAD)

DETAILED DESCRIPTION:
To evaluate the improvement of the quality of life of antidepressant monotherapy on Chinese patients who meet DSM-5 criteria for the comorbidity of MDD and GAD. To monitor adverse events (AEs) and serious adverse events (SAEs) of antidepressant monotherapy

ELIGIBILITY:
Inclusion Criteria:

1. First episode outpatients in department of psychiatry, aged 18-65 years
2. Comorbidity of MDD and GAD according to DSM-5 criteria Hamilton Depression score (HAMD) of ≥18 at screening
3. HAMA≥14 at screening
4. Medically stable
5. Provision of written, informed consent.

Exclusion Criteria:

1. Suicide ideation
2. Use antidepressants within at least 14 days before study begin
3. Substance or alcohol dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence)
4. Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse within 4 weeks prior to enrolment
5. Unstable or inadequately treated medical illness (e.g. congestive heart failure, angina pectoris, hypertension, renal or hepatic dysfunction, cerebrovascular disease ) as judged by the investigator
6. Women in pregnancy or lactation
7. Medical conditions that would affect absorption, distribution, metabolism or excretion of study treatment.
8. Medical history with seizure disorder, except for febrile convulsion
9. Participation in another clinical study within 4 weeks (or longer time according to the local requirement)
10. Receive Electroconvulsive therapy (ECT) before study begin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients who meet DSM-5 criteria for the combidity of MDD and GAD
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-01 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the score of HAMD17 (Hamilton Depression Rating Scale) and HAMA (Hamilton Anxiety Rating Scale) of patients in each time between two groups | one year
  The efficacy variables is include:
  Onset rate: proportion of patient with at least 20% reduction in HAMD total score after 1 week Response rate: proportion of patient with at least 50% reduction in HAMD total score Remission rate: remission is defined as HAMD ≤ 7; remission rate is proportion of patients with remission HAMD total score change from baseline to week 6 and to week 24 (LOCF) during the study.
  HAMA and the Mos36-item Short Form Health Survey (SF-36) score Change from baseline to week6 and to week 24 (LOCF) during the study.

SECONDARY OUTCOMES:
Evaluate the symptom of depression, anxiety and quality of life in each time between two groups | one year

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Huang, MD, Principal Investigator — Fudan University; Jian l Ji, MD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China